CLINICAL TRIAL: NCT06391697
Title: A Feasibility Study Evaluating the Magnetic Bead Tracking System and Its Safety and Efficacy When Used With the e-OPRA Implant System and a Bionic External Prosthesis to Improve Prosthetic Controllability for Persons With Transtibial Amputation
Brief Title: Magnetic Bead Tracking System and eOPRA Implant System With Bionic Prosthesis for Transtibial Amputees
Acronym: TTeOPRA+MB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (MIT) (Unknown); Integrum (Industry)
Responsible Party: Principal Investigator, Matthew Carty, Roberta and Stephen R. Weiner Distinguished Chair in Surgery, Staff Surgeon BWH, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024P00006
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Amputation
Keywords: prosthesis; osseointegration; neural transmission; magnetic beads

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- eOPRA Implant System for Transtibial Amputees and Magnetic Bead Tracking System (Experimental): Implantation of e-OPRA Implant System and Magnetic Bead Tracking System in lower limb.
  Interventions: Device: eOPRA Implant System for Transtibial Amputees and Magnetic Bead Tracking System

INTERVENTIONS:
Device: eOPRA Implant System for Transtibial Amputees and Magnetic Bead Tracking System — The Magnetic Bead Tracking System is an investigational device that consists of pairs of magnetic beads, and a set of magnetic field sensors that measure and track the length of muscles and the speed at which they move in real-time. When the beads are implanted in muscle in the residual limb of an amputee, the muscle length signal is communicated to an investigational, robotic ankle-foot prosthesis.
  The e-OPRA is an investigational implant system that lets a lower leg prosthesis attach securely to the remaining tibia bone. The e-OPRA device has been designed so that it can be implanted with an electrode set that consists of an electrical connector and electrodes to allow it to be used with both a neuro-mechanical (powered) prosthesis system, in addition to the standard prosthesis.
  The operation to implant these devices will represent a modification of the surgical technique currently employed for standard below knee amputation.
  Other Names: eOPRA; e-Osseointegrated Prosthesis for the Rehabilitation of Amputees

SUMMARY:
The e-OPRA Implant System, is a further development of the OPRA (Osseointegrated Prostheses for the Rehabilitation of Amputees) Implant System. The e-OPRA Implant system is an implant system for direct skeletal anchorage of amputation prostheses. The added feature in the e-OPRA Implant system, is a bidirectional interface into the human body that allows permanent and reliable communication using implanted electrodes. These electrodes will provide long-term stable bioelectric signals for an improved control of the prosthetic limb. The Magnetic Bead Tracking System, which will be implanted and used in combination with the e-OPRA Implant system, is an investigational device that consists of pairs of magnetic beads, and a set of magnetic field sensors that measure and track the length of muscles and the speed at which they move in real-time. When the beads are implanted in muscle in the residual limb of an amputee, the muscle length signal is communicated to an investigational, robotic ankle-foot prosthesis. The purpose of the study is to evaluate the feasibility of a transtibial amputee with the e-OPRA Implant System and Magnetic Bead Tracking System exhibiting full neural control over a neuro-mechanical prosthetic system.

A maximum of seven subjects will be enrolled. Each subject will undergo one or more surgeries where the e-OPRA Implant System and Magnetic Bead Tracking System will be implanted. The subjects will participate in follow-up sessions the last of which occurs approximately 24 months after the surgery. This is a prospective, non-randomized, uncontrolled study.

DETAILED DESCRIPTION:
Normalization of function for individuals with limb amputation is within reach, and will be achieved by smart implants capable of bi-directional communication between brain and machine via bone-anchored, interactive, powered prosthetic components. Rehabilitation of patients with expected high physical activity level, such as after amputation due to trauma or cancer, is currently limited by dependence on an external socket for the mechanical attachment of the prosthesis to the residuum. Despite the use of advanced materials and fabrication methods, socket interfaces routinely cause sores, chafing, pain, increased energy expenditure, and a decreased quality of life. Novel surgical techniques using osseointegrated transdermal titanium implants, now validated in Europe for over 25 years, obviate the need for painful sockets by establishing a direct, load-bearing link between skeleton and prosthesis. This system also promises a transformative breakthrough in neuroprosthetics, because it allows for fully internal, high bandwidth, stable neural connections. In a paper recently published in Science Translational Medicine, implanted muscle and nerve cuff electrodes were added to the osseointegrated device, creating a bi- directional efferent-afferent interface utilizing a safe and immune-sealed osseo-conduit. Commenting on this work, the editor stated, "Osseointegration could revolutionize the field of neuroprosthetics, giving patients more intuitive control and more freedom of movement."

Investigators have sought to advance bionic prostheses with sufficient degrees of freedom for performing natural tasks, such as manipulating objects in the case of upper-extremity prostheses, or walking and running for lower-extremity systems. Nonetheless, afferent feedback has not played a major role in any clinically-viable amputation prostheses, despite being critical for biomimetic control. This deficiency can, in large part, be attributed to a lack of clinically-available methodologies for sustained communication with the peripheral nervous system. There is no existing platform capable of invasive, robust, and permanent communication with the peripheral nervous system in a high-demand clinical set- ting. Only by bringing together critical technologies and expertise will it be possible to create a bionic limb replacement system with adequate suspension, load transmission, motor control, proprioceptive feedback, and external mechatronics that resemble the mass, volume and dynamics of the missing biological limb.

To develop the most advanced clinically- viable artificial limb and achieve the next level of prosthetic technology integration, a multi-disciplinary scientific team has been assembled with members from Massachusetts Institute of Technology (MIT: Carty, Herr, Brånemark) and Brigham and Women's Hospital (BWH: Carty, Ferrone). With proprioceptive afferent feedback, we seek to demonstrate that a person with transtibial amputation can exhibit full volitional control over a neuro-mechanical prosthetic system where key walking metrics are normalized, including preferred speed, metabolism and joint dynamics. It is the view of the proposers that the scope of this research is fundamental wherein the results will be shared broadly within the scientific community.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 22-65 at the time of surgery.
2. The subject must already have been implanted with the e-OPRA Implant System at the transtibial level or must have an existing unilateral or bilateral transtibial amputation or a medical condition requiring performance of a unilateral or bilateral transtibial amputation with a minimum of 8 cm of residual tibia after amputation, such that the subject will be implanted with the e-OPRA Implant System. (OPTION 1)
3. If the subject does not already have the e-OPRA Implant System, the subject must have undergone independent consultation with at least two lower extremity surgical specialists to ensure they have exhausted all limb salvage options prior to undergoing amputation, as well as a psychiatric evaluation to ensure appropriate capacity and volition. (OPTION 2)
4. The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above, as confirmed by study investigators).
5. The patient must have adequate soft tissue bulk and muscle mass present in the operative limb to support appropriate wound healing.
6. In the opinion of the investigator, normal cognitive function and absence of any physical limitations, addictive diseases or underlying medical conditions that may preclude the patient from being a good study candidate.
7. Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.
8. Willingness and ability to provide informed consent to participate in the study.

Exclusion Criteria:

1. Subjects with any active skin disease in the tested limb.
2. Subjects with severe co morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life. expectancy, vulnerable patient population, BMI >40, etc.).
3. For subjects who have not yet been implanted with the e-OPRA Implant System, subjects who would have less than 2 mm of remaining cortex bone available around the implant, if implanted.
4. Subjects with advanced atrophic muscle and/or compromised soft tissue coverage in the operative limb.
5. Subjects with evidence of or a documented history of severe peripheral vascular disease, diabetes mellitus (type I or type II), skin diseases, neuropathy or neuropathic disease and severe phantom pain, or osteoporosis, such that, in the opinion of the investigator, will not allow the subject to be a good study candidate.
6. Subjects with a history of systemically administered corticosteroids, immune-suppressive therapy or chemotherapy drugs within six (6) months of implant surgery.
7. Subjects with a known need of future MRIs.
8. Subjects currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study.
9. Active smokers will be excluded from candidacy; those patients willing to undergo tobacco cessation will need to be completely abstinent from tobacco use for at least 6 weeks preoperatively.
10. Women who are pregnant, lactating or planning a pregnancy during the first twelve (12) months of the post-surgical follow-up.
11. Subject has an allergy to any component of the device.
12. Concurrent illness, disability or geographical residence would hamper attendance at required study visits.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
number of participants out of total who undergo device implantation (aim: 7 participants) who can complete robotics testing activities | 3 - 24 months postop for all study participants
  testing activities include subject stability assessments, free space control activities using EMG, bead migration assessments, walking gait assessments and single-leg balance assessments
number of participants out of total who undergo device implantation (aim: 7 participants) who still have device successfully implanted at 24 months postop | 24 months postop for all study participants
  successful implantation at 24 months is defined as having both eOPRA Implant System and Magnetic Beads Tracking System intact with no plans for removal due to device-related safety concern

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carty, MD, Principal Investigator — Brigham and Women's Hospital; Hugh Herr, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - MIT Media Lab, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No